CLINICAL TRIAL: NCT06650644
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Investigator-initiated Human Study to Evaluate the Efficacy and Safety of Lactococcus Lactis KD10 Powder in Improving Autism Spectrum Symptoms in Pediatric Patients With Autism Spectrum Disorder.
Brief Title: A Study to Evaluate the Efficacy and Safety of Lactococcus Lactis KD10 Powder for Improving Autism Spectrum Symptoms in Children With Autism Spectrum Symptoms.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miae Oh (Other)
Collaborators: KoBioLabs (Industry); Korea University (Other)
Responsible Party: Sponsor-Investigator, Miae Oh, Professor, Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD10; 20023378 (Other Grant/Funding Number: The Ministry of Trade, Industry and Energy(MOTIE, Korea))
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Lactococcus lactis; Human Study
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test food group (Experimental): Food name: Lactococcus lactis KD10
  Interventions: Dietary Supplement: Lactococcus lactis KD10 (health food)
- Control food group (Placebo Comparator): Food name: Placebo of Lactococcus lactis KD10
  Interventions: Other: Placebo of Lactococcus lactis KD10

INTERVENTIONS:
Other: Placebo of Lactococcus lactis KD10 — * Food Name: Placebo of Lactococcus lactis KD10
  * Ingredients: Natural pigment enteric-coated granules preparation
  * Appearance and Formulation: Granules/Powder
  * Dosage/Amount: 1 pack once a day
  * Dosage period and route: Oral intake of 1 pack once a day for 12 weeks 30 minutes after meals
  Arms: Control food group
Dietary Supplement: Lactococcus lactis KD10 (health food) — * Food Name: Lactococcus lactis KD10 (health food)
  * Ingredients: Freeze-dried Lactococcus lactis enteric-coated granules preparation
  * Appearance and Formulation: Granules/Powder
  * Dosage/Amount: 1 pack once a day
  * Administration Period and Route: Oral intake of 1 pack once a day for 12 weeks 30 minutes after meals
  Arms: Test food group

SUMMARY:
This human study aims to evaluate the efficacy and safety of Lactococcus lactis KD10 powder for improving autism spectrum disorder symptoms in patients with autism spectrum disorder.

DETAILED DESCRIPTION:
The purpose of this human study is to confirm the change rate (%) in the main symptoms of autism spectrum disorder after 12 weeks of taking Lactococcus lactis KD10 powder in subjects with autism spectrum disorder.

In addition, we will conduct tests using various evaluation scales at the 12-week point to evaluate the degree of autism spectrum disorder symptoms and coexisting disease symptoms, and to evaluate the overall safety during the human study period.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 years or older and 7 years and 7 months or younger
2. Those diagnosed with autism spectrum disorder through a standardized diagnostic tool according to the diagnostic criteria for autism spectrum disorder in the DSM-5 (Diagnostic and Statistical Manual of Mental disorder-5) at the time of screening [Diagnostic tool: Korean version of Autism Diagnostic Observation Schedule version 2 (K-ADOS-2), Korean version of Autism Diagnostic Interview-Revised (K-ADI-R)] (However, if diagnosed with autism spectrum disorder through a diagnostic evaluation within 6 months of screening, only the K-ADOS-2 test will be re-evaluated.)
3. Those judged by the investigator on the day of screening to be able to consume the food for this human test (control food) without chewing it, with water or the provided puree
4. Those subjects or/and their legal representatives who voluntarily agreed to participate in this human test and signed a written consent form and a consent form for research on human-derived materials
5. A person who can provide reliable information on the condition of the test subject during the human test period, attend all planned visits to the institution, supervise the intake of food for human test, and have the participation of a parent or the same legal representative who can fully understand and speak Korean, and conduct a questionnaire evaluation of the subject.

Exclusion Criteria:

[Screening Visit (Visit 1)]

1. Those with the following medical history, concomitant diseases, or surgical history at the time of screening ① Severe psychosis that may affect this test other than autism spectrum disorder

   ② History of organic brain disease, neurological disorder, uncontrolled epilepsy, or seizures. However, simple febrile seizures can be included at the investigator's discretion

   ③ Genetic diseases (Rett syndrome, Down syndrome, Fragile X syndrome, etc.) However, participation is allowed at the investigator's discretion only if it is confirmed to be a genetic disease that does not affect the results of this test

   ④ Gastrointestinal diseases and surgical history that may affect the intestinal absorption of food for human testing (simple appendectomy, hernia surgery are allowed)

   ⑤ Those with sensory abnormalities such as congenital hearing loss
2. Those with uncontrolled medical conditions (including arrhythmia, cancer, severe heart/kidney disease) during the screening period
3. Those who exhibit serious self-harming or other-harming behaviors that require medical treatment at the investigator's discretion during the screening period
4. Those who have been confirmed to have taken the following drugs within 2 weeks prior to screening or are expected to take the following drugs during the human application test period. However, for drugs with a sufficient washout period exceeding 2 weeks, a washout period of at least 5 times the maximum half-life must be confirmed before the screening time.

   ① Antipsychotic drugs (antipsychotic, psychostimulant, antidepressant, anxiolytic, mood stabilizer, and neuroleptic agents). If there is no change in the type or dosage of the drug within 3 months of screening due to long-term use, participation is possible at the investigator's discretion

   ② Selective Serotonin Reuptake Inhibitor (SSRI)
5. Those with the following test results confirmed during screening

   ① Moderate or higher renal impairment (eGFR <60mL/min/1.73m2)

   ② Moderate or higher hepatic impairment(AST or ALT >3 x ULN)
6. Those who cannot receive intravenous injection for blood collection
7. Those who have difficulty consuming human application test food or are sensitive or allergic to human test food
8. Those who participated in other clinical trials or human trials within 4 weeks prior to screening and were administered or consumed clinical trial drugs or human test food or were applied with clinical trial medical devices
9. Those who are judged unsuitable for participation in human trials by the investigator

[baseline visit (Visit 2)]

1. Those with unsuitable items when reconfirming the selection/exclusion criteria at the time of randomization
2. Those judged unsuitable for participation in this human study by the investigator other than the above

Ages: 36 Months to 91 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Change rate of major symptoms of autism spectrum disorder (%)_Korean version of Vineland Adaptive Behavior Scale-II(K-VABS-II) | Baseline(0 weeks), 12 weeks
  To determine the change rate (%) in major symptoms of autism spectrum disorder

SECONDARY OUTCOMES:
Social Skills Change Rate (%)_Korean version of Autism Diagnostic Observation Schedule version 2(K-ADOS-2) | Baseline(0 weeks), 12 weeks
  To observe and diagnose patients with autism spectrum disorder.
Social Skills Change Rate (%)_Korean version of Childhood Autism Rating Scale-2(K-CARS-2) | Baseline(0 weeks), 12 weeks
  Developmental screening for children and adolescents suspected of having autism spectrum disorder
Social Skills Change Rate (%)_Social Responsiveness Scale-2(SRS-2) | Baseline(0 weeks), 12 weeks
  A questionnaire asking about the characteristics of children's social interactions.
Social Skills Change Rate (%)_Korean version of Social Communication Questionnaire(K-SCQ) | Baseline(0 weeks), 12 weeks
  Questions to screen for Autism Spectrum Disorder.
Social Skills Change Rate (%)_Aberrant Behavior Checklist-II | Baseline(0 weeks), 12 weeks
  Symptom checklist to assess problem behaviors in children with developmental disabilities.
Level of functioning Change Rate (%)_Korean version of Wechsler Primary and Preschool Scale Intelligence-Ⅳ(K-WPPSI-Ⅳ) | Baseline(0 weeks), 12 weeks
  Assess cognitive abilities
Level of functioning Change Rate (%)_CGI-S (Clinical Global Impression-Severity) | Baseline(0 weeks), 12 weeks
  CGI-S is a scale that clinicians use to objectively measure the overall severity of a disease.
Level of functioning Change Rate (%)_CGI-I (Clinical Global Impression-Improvement) | 12 weeks
  CGI-I is an assessment that evaluates whether the patient has improved or worsened after a therapeutic intervention compared to before the intervention.
Executive function Change Rate (%)_Children's Color Trail making Test 1&2(CCTT 1&2) | Baseline(0 weeks), 12 weeks
  It is a neuropsychological test tool that evaluates cognitive function and can also evaluate attention and executive functions.
Executive function Change Rate (%)_Stroop Test (Color & word) | Baseline(0 weeks), 12 weeks
  Measures attention and response inhibition.
Executive function Change Rate (%)_ Advanced Test of Attention(ATA) | Baseline(0 weeks), 12 weeks
  A precise attention test program that measures sustained and selective attention and impulse control.
Executive function Change Rate (%)_Korean version of ADHD Rating Scale-IV(K-ARS-4) | Baseline(0 weeks), 12 weeks
  Assessing ADHD symptoms in school-aged children.
Sleep disturbance Change Rate (%)_The Korean version of the Children's Sleep Habits Questionnaire | Baseline(0 weeks), 12 weeks
  Assess overall sleep habits, including sleep behaviors, sleep problems, and sleep disorders in school-aged children.
Anxiety Change Rate (%)_Korean version of Child Behavior Checklist (K-CBCL) | Baseline(0 weeks), 12 weeks
  A scale for examining emotional and behavioral problems in children with autism spectrum disorder.
Anxiety Change Rate (%)_Korean form of the State and Trait Anxiety Inventory for Children (K-STAIC) | Baseline(0 weeks), 12 weeks
  Assessment tool to measure anxiety in children.
GI trouble Change Rate (%)_Profile Of Toileting Issue (POTI) | Baseline(0 weeks), 12 weeks
  A scale to check toilet use problems.
Sensory Change Rate (%)_Short Sensory Profile-2 (SSP-2) | Baseline(0 weeks), 12 weeks
  Measuring children's responses to sensory processing in everyday life.
Parenting stress change rate (%)_Korean version of Parenting Stress Index Forth edition-Short Form (K-PSI-4-SF) | Baseline(0 weeks), 12 weeks
  Parenting Stress Measurement Tool

OTHER OUTCOMES:
Rate of change in the type and number of intestinal flora etc. through fecal collection and fecal flora analysis (%) | Baseline(0 weeks), 12 weeks
  <Exploratory endpoint> Using stool collection container and DNA stabilization kit containers, we would like to determine the overall changes by flora-intestinal(Type, number etc.) by fecal flora analysis (%).
Rate of change in blood biomarker values | Screening visit (-4 weeks) or Baseline(0 weeks), 12 weeks
  <Exploratory endpoint> we seek to explore the association between autism and blood biomarkers.
Blood collection for DNA analysis | Screening visit (-4 weeks) or Baseline(0 weeks)
  <Exploratory endpoint> DNA Identification of Subjects with Autism Spectrum Disorder.
Collecting and analyzing information on microorganisms (DNA type, etc.) in the oral cavity by collecting oral samples (such as saliva) | Screening visit (-4 weeks) or Baseline(0 weeks), 12 weeks
  <Exploratory endpoint> The purpose of this outcome is to explore the types of microbiomes identified etc. in the oral cavity of subjects with autism spectrum disorder.
  This outcome will be conducted twice (Visit 1 or Visit 2, Visit 4) using the AccuBuccal Collection kit. AccuBuccal Collection kits, they will be collected by the investigator, who will use the kit provided to collect samples.
  Subjects should refrain from brushing their teeth, washing their tongue, and eating coffee, beverages, water, and food at least two hours before collection.

CONTACTS AND LOCATIONS:
Overall Officials: Miae OH, Principal Investigator — Kyunghee University Medical Center
Locations (2):
- South Korea (2):
  - Seoul national University buseoul national University bundang hospitalndang hospital, Seongnam-si, Gyeonggi-do
  - Kyung Hee University Medical Center, Seoul, Kyungheedae-ro, Dongdaemun-gu

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share any related individual participant data within reasonable request which can be obtained from the principal investigators.